CLINICAL TRIAL: NCT03055897
Title: Tear Film Innovations iLux Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tear Film Innovations, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2020-11

CONDITIONS: Meibomian Gland Dysfunction; Evaporative Dry Eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- iLux 2020 System (Experimental): Meibomian gland treatment (Day 0) according to instructions for use (IFU)/User Manual
  Interventions: Device: iLux 2020 System

INTERVENTIONS:
Device: iLux 2020 System — Medical device that applies localized heat and pressure therapy to the eyelid in order to express melted meibum from obstructed glands

SUMMARY:
The objective of this study was to measure the temperature of the cornea and surrounding eye tissue temperature immediately after heating the eyelids with the iLux device using the protocol treatment profile. Eligible participants attended one treatment visit, with follow-up one day following the procedure.

DETAILED DESCRIPTION:
Alcon Research, LLC, acquired TearFilm Innovations, Inc., in December 2018. This study was designed and conducted by TearFilm Innovations, Inc. The study results were collected, analyzed, and provided by TearFilm Innovations, Inc., to Alcon Research, LLC.

ELIGIBILITY:
Key Inclusion Criteria:

- Sign written informed consent prior to study participation

Key Exclusion Criteria:

* History of ocular surgery within 1 year
* Active ocular infection
* Ocular surface abnormality; lid surface abnormalities
* Pregnant, nursing or not utilizing adequate birth control measures
* Other protocol-specified exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2016-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. CDMA Project Lead, CDMA Ocular Health, Study Director — Alcon Research, LLC
Locations (1):
- TearFilm Innovations Investigative Site, Encinitas, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one investigative site located in the United States.
Pre-assignment Details: This reporting group includes all enrolled participants.
Period: Overall Study
Arm/Group | iLux 2020 System
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | iLux 2020 System
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (15.1)
Sex/Gender, Customized [Number; unit: participants]
  Male | 7
  Not reported | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 1
  White | 11
  Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Overall Maximum Temperature of the Cornea and Surrounding Eye Tissue Immediately Post-treatment
Description: Post-heating values were obtained by infrared camera for each participant. The cornea, the eyelid, and the surface tissue surrounding the eye were measured. Both eyes contributed to the analysis. No formal hypothesis testing was specified.
Time Frame: Day 0 immediately post-treatment
Population: Safety Analysis Set: All subjects enrolled and treated
Measure: Mean (Standard Deviation); unit: degrees Celsius
Units Other Than Participants: eyes
Arm/Group | iLux 2020 System
Number analyzed (Participants) | 15
Number analyzed (eyes) | 30
degrees Celsius
  Corneal temperature | 37.7 (0.5)
  Eyelid temperature | 38.5 (0.8)
  Surface temperature | 38.2 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant from time of enrollment until time of study exit, approximately 2 days.
Description: An adverse event was defined as any untoward and unintended sign, symptom or disease temporally associated with the use of an investigational drug or device, or other protocol-imposed intervention, regardless of the suspected cause. All participants exposed to the study treatment were evaluated for adverse events.
Arm/Group | iLux 2020 System
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT03055897/Prot_SAP_000.pdf